CLINICAL TRIAL: NCT04264962
Title: Yang Yin Fu Zheng Jie Du Therapy in Recurrence of Hepatocellular Carcinoma Less Than 3 cm in Diameter
Acronym: YYFZJDTRHCLT3D
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Ditan Hospital (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhiyun Yang, Archiater, Professor, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingDHYZY
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yang Yin Fu Zheng Jie Du therapy (Experimental)
  Interventions: Drug: Yang Yin Fu Zheng Jie Du therapy; Other: Routine medical care
- Routine medical care (Placebo Comparator)
  Interventions: Other: Routine medical care

INTERVENTIONS:
Drug: Yang Yin Fu Zheng Jie Du therapy — Yang Yin Fu Zheng Jie Du is a Chinese herbal compound.
  Arms: Yang Yin Fu Zheng Jie Du therapy
Other: Routine medical care — Routine medical care

SUMMARY:
Clinical research of Yang Yin Fu Zheng Jie Du therapy in recurrence of Hepatocellular Carcinoma less than 3 cm in diameter.The purpose of this study is to observe the efficacy of routine medical care combined with Yang Yin Fu Zheng Jie Du therapy in 1 year recurrence for patients belong to Hepatocellular Carcinoma less than 3 cm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of hepatocellular carcinoma
* Ages Eligible for Study: ≤75 years old;
* The size of the main nodule and multi-centricity (single lesion, three nodules ≤3 cm)
* After transarterial chemoembolisation (TACE) or radiofrequency ablation (RFA)
* Surgery cannot be allowed;
* Informed consent from the patient.

Exclusion Criteria:

* Serious problem of heart, lung, or kidney with severe dysfunction;
* Pregnant or child breast feeding women;
* Mental or cognitive disorders;
* Participating in other drug trials;
* Who are allergic to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Recurrance rate | 1 year

SECONDARY OUTCOMES:
Objective response rate | 1 year
quality of life (QOL) questionnaire | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiyun Yang, Beijing, Beijing Municipality, China